CLINICAL TRIAL: NCT03507439
Title: Real Life Multimarker Monitoring in Patients With Heart Failure
Brief Title: REALIsM-HF Pilot Study
Acronym: REALIsM-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19167
Record Dates: First submitted 2018-04-20; First posted 2018-04-25 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2022-07

CONDITIONS: Heart Failure
Keywords: Heart failure with preserved ejection fraction (HFpEF); Heart failure with reduced ejection fraction (HFrEF)
MeSH Terms: conditions — Heart Failure | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- HFrEF (Experimental): Participants with established diagnosis of heart failure with reduced ejection fraction (HFrEF; EF ≤ 35%) wore the AVIVO MPM System or VitalPatch biosensor for 5 monitoring periods with patches applied on Day 0, 9, 16, 77 and 84; and the DynaPort Move Monitor belt for 2 monitoring periods with belts applied on Day 9 and Day 77.
  Interventions: Device: AVIVO Mobile Patient Management (MPM) System; Device: VitalPatch biosensor; Device: DynaPort Move Monitor
- HFpEF (Experimental): Participants with established diagnosis of heart failure with preserved ejection fraction (HFpEF; EF ≥ 45%) wore the AVIVO MPM System or VitalPatch biosensor for 5 monitoring periods with patches applied on Day 0, 9, 16, 77 and 84; and the DynaPort Move Monitor belt for 2 monitoring periods with belts applied on Day 9 and Day 77.
  Interventions: Device: AVIVO Mobile Patient Management (MPM) System; Device: VitalPatch biosensor; Device: DynaPort Move Monitor

INTERVENTIONS:
Device: AVIVO Mobile Patient Management (MPM) System — Wearable, wireless physiological monitoring and arrhythmia detection system, used by participants for 5 monitoring periods of 5 days each in the study
Device: VitalPatch biosensor — Wearable, wireless physiological monitoring and arrhythmia detection system, used by participants for 5 monitoring periods of 5 days each in the study
Device: DynaPort Move Monitor — Wearable device for ambulatory monitoring of physical activity, used by participants for 2 monitoring periods of 7 days each in the study

SUMMARY:
The study aims to explore two marketed devices providing a multimarker monitoring including physical activity under real-life conditions in patients with heart failure with preserved ejection fraction (HFpEF) and with heart failure and reduced ejection fraction (HFrEF). It aims to identify potential novel endpoints for future heart failure trials by exploring clinically relevant changes over time and correlations/associations with conventional endpoints such as the six minute walking distance (6MWD), biomarkers and clinical events. Furthermore, it aims to address the challenges and feasibility of implementing device based measurements under real-life conditions.

DETAILED DESCRIPTION:
Device 1 AVIVO Mobile Patient Management System (Medtronic USA), substituted by VitalPatch biosensor (VitalConnect USA) during the course of the study Device 2 DynaPort Move Monitor (McRoberts, NL)

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed before any study-specific procedure
* Men or women aged 45 years and older
* Established diagnosis of chronic heart failure NYHA class II-IV
* Worsening heart failure requiring hospitalization for the initiation of intensification of heart failure therapy with at least one of the following: a) BNP ≥ 100 pg/mL or NT-proBNP ≥ 400 pg/mL (sinus rhythm) OR BNP ≥ 300 pg/mL or NT-proBNP ≥ 1200 pg/mL (atrial fibrillation); OR b) Radiographic evidence of pulmonary congestion (interstitial edema, pulmonary venous hypertension, vascular congestion, pleural effusion); OR c) Catheterization documented elevated filling pressures at rest (left ventricular end-diastolic pressure ≥15 mmHg or pulmonary capillary wedge pressure ≥ 20 mmHg) or with exercise (pulmonary capillary wedge pressure ≥ 25 mmHg) OR Ambulatory patients with a history of heart failure on individually optimized treatment with HF medications unless contraindicated or not tolerated, for at least 12 weeks and at least one of the following: a) Hospitalization for heart failure within the past 12 months; OR b) BNP ≥ 100 pg/mL or NT-proBNP ≥ 400 pg/mL (sinus rhythm) or BNP ≥ 300 pg/mL or NT-proBNP ≥ 1200 pg/mL (atrial fibrillation)
* For HFrEF only: EF ≤35% assessed by any imaging modality (e.g. echocardiography, cardiac magnetic resonance, cine levocardiography) within 12 months prior to study inclusion
* For HFpEF only: EF ≥45% assessed by any imaging modality (e.g. echocardiography, cardiac magnetic resonance, cine levocardiography) within 12 months prior to study inclusion
* Willingness to wear the DynaPort Move Monitor accelerometer belt and VitalPatch Biosensor during the trial
* Body size allows wearing of the accelerometer belt as confirmed by ability to comfortably fasten the test belt provided for the screening process

Exclusion Criteria

* Inability to comply with planned study procedures or to comply with study protocol requirements; this includes completing required data collection, and attending required follow up study visits
* Hemoglobin < 8.0 g/dl
* Acute coronary syndrome or percutaneous coronary intervention within 3 months prior to informed consent
* Listing for heart transplantation and / or anticipated implantation of a ventricular assist device
* Inability to exercise: wheelchair / scooter / walker dependent; dependent on supplemental oxygen
* Known clinically significant persistent coronary ischemia (based on medical history, a preexisting or a recent clinical stress test)
* HF is not the primary factor limiting activity within the last three months as indicated by the patient affirming #1, #2 or #3 of the following questionnaire: My ability to be active is most limited by: #1 - Joint, foot, leg, hip or back pain; #2 - Unsteadiness or dizziness impairing daily mobility; #3 - Lifestyle, weather, or I just don't like to be active
* Occurrence of any of the following within 3 months prior to informed consent: Myocardial infarction, Hospitalization for unstable angina, Stroke or transient ischemic attack, Coronary artery bypass graft (CABG), Percutaneous coronary intervention (PCI), Implantation of a cardiac resynchronization therapy device (CRTD), Major surgery (that could interfere with patients' ability to exercise)
* PCI, CABG or implantation of a CRTD planned between randomization and Visit 4
* Subject who cannot tolerate placement of external patch monitor on chest in the proposed location (ECG lead II orientation)
* Subject with known allergies or hypersensitivities to adhesives or hydrogels
* Severe uncorrected valvular heart disease
* Known clinically relevant ventricular arrhythmias (sustained ventricular tachycardia, ventricular flutter or fibrillation)
* Severe pulmonary disease with any of the following: Requirement of continuous (home) oxygen or History of chronic obstructive pulmonary disease ≥ GOLD III
* Previous (within 30 days or 5 half-lives of the investigational drug, whichever is longer) or concomitant participation in another clinical study with investigational medicinal product(s) or device(s)
* Any condition or therapy, which would make the patient unsuitable for the study, or life expectancy less than 12 months (e.g. active malignancy)
* Heavy alcohol consumption or the use of illicit drugs that, in the opinion of the investigator, may interfere with the patient's safety and / or compliance
* Patients who regularly (> 1x per week) swim, do water aerobics or go to the sauna, unwilling to omit this activity while needing to wear the study specific medical devices
* Active myocarditis
* Primary hypertrophic cardiomyopathy
* Constrictive pericarditis or pericardial tamponade
* Close affiliation with the investigational site, e.g. a close relative of the investigator, dependent person (e.g. employee or student of the investigational site)
* Previous participate in the study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-03-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States
- Germany (3):
  - Universitätsklinikum Köln, Cologne, North Rhine-Westphalia
  - Heinrich-Heine-Universität Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Charité - Campus Virchow-Klinikum (CVK), Berlin
- ASST Spedali Civili di Brescia, Brescia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at multiple centers in 3 countries between 06 APR 2018 (first participant first visit) and 12 MAR 2021 (last participant last visit).
Pre-assignment Details: Overall, 29 participants were screened, of which 2 participants were screening failures and 27 participants received at least one device.
Period: Overall Study
Arm/Group | HFrEF | HFpEF
Started | 14 | 13
Completed | 10 | 11
Not Completed | 4 | 2
Not completed — Other | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) : all participants that were enrolled into the study and that wore at least one device
Groups:
- Total: Total of all reporting groups
Arm/Group | HFrEF | HFpEF | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.7 (9.2) | 73.8 (8.9) | 69.1 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 7
  Male | 13 | 7 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
6-minute walking distance (6MWD) [Mean (Full Range); unit: Meters (m)] — 6-minute walking distance (6MWD) is a exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. An increase in the distance walked indicates improvement in basic mobility. Population: Participants in full analysis set (FAS) with evaluable data for this evaluation
  Meters (m)
    number analyzed (Participants) | 12 | 12 | 24
    (all) | 382 [253 to 575] | 291 [92 to 506] | 337 [92 to 575]
Quality of Life as measured by the Kansas City Cardiomyopathy Questionnaire score [Median (Full Range); unit: Scores on a scale] — The Kansas City Cardiomyopathy Questionnaire (KCCQ) is the leading health-related quality-of-life measure for patients with heart failure (HF). Physical Limitation ranges 0-100. Total Symptom Score (range 0-100) combines the Symptom Frequency and the Symptom Burden scores; Clinical Summary Score (range 0-100) combines the Total Symptom and Physical Limitation scores to replicate the NYHA classification; Overall Summary Score (range 0-100) includes the Total Symptom, Physical Limitation, Social Limitations, and Quality of Life scores. Higher scores indicate more favorable states. Population: Participants in full analysis set (FAS) with evaluable data for this evaluation
  Scores on a scale
    Total Symptom Score: number analyzed (Participants) | 7 | 7 | 14
    Total Symptom Score | 64.0 [53 to 100] | 33.0 [4 to 100] | 61.0 [4 to 100]
    Clinical Summary Score: number analyzed (Participants) | 7 | 7 | 14
    Clinical Summary Score | 68.0 [37 to 98] | 41.0 [8 to 83] | 66.0 [8 to 98]
    Overall Summary Score: number analyzed (Participants) | 7 | 7 | 14
    Overall Summary Score | 67.0 [29 to 96] | 43.0 [8 to 81] | 64.5 [8 to 96]
    Physical Limitation Score: number analyzed (Participants) | 7 | 7 | 14
    Physical Limitation Score | 71.0 [21 to 96] | 54.0 [8 to 75] | 65.0 [8 to 96]
Copeptin [Mean (Standard Deviation); unit: Picomoles per litre (pmol/L)] — Biomarkers were determined in plasma/serum by a central laboratory using validated assays platforms including appropriate quality controls. Population: Participants in full analysis set (FAS) with evaluable data for this evaluation
  Picomoles per litre (pmol/L)
    number analyzed (Participants) | 9 | 8 | 17
    (all) | 47.047 (37.744) | 31.551 (23.693) | 39.755 (31.960)
Galectin-3 [Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)] — Biomarkers were determined in plasma/serum by a central laboratory using validated assays platforms including appropriate quality controls. Population: Participants in full analysis set (FAS) with evaluable data for this evaluation
  Nanograms per milliliter (ng/mL)
    number analyzed (Participants) | 9 | 8 | 17
    (all) | 15.622 (9.403) | 12.265 (4.988) | 14.042 (7.621)
Growth differentiation factor 15 (GDF 15) [Mean (Standard Deviation); unit: Picograms per millilitre (pg/mL)] — Biomarkers were determined in plasma/serum by a central laboratory using validated assays platforms including appropriate quality controls. Population: Participants in full analysis set (FAS) with evaluable data for this evaluation
  Picograms per millilitre (pg/mL)
    number analyzed (Participants) | 9 | 8 | 17
    (all) | 4740.2 (4840.0) | 2689.6 (1512.6) | 3775.2 (3718.5)
Human interleukin-1 Receptor 4 / ST2 [Mean (Standard Deviation); unit: Picograms per litre (pg/L)] — Biomarkers were determined in plasma/serum by a central laboratory using validated assays platforms including appropriate quality controls. Population: Participants in full analysis set (FAS) with evaluable data for this evaluation
  Picograms per litre (pg/L)
    number analyzed (Participants) | 9 | 8 | 17
    (all) | 35.09 (14.33) | 28.69 (18.45) | 32.08 (16.20)
Human Insulin-like Growth Factor Binding [Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)] — Biomarkers were determined in plasma/serum by a central laboratory using validated assays platforms including appropriate quality controls. Population: Participants in full analysis set (FAS) with evaluable data for this evaluation
  Nanograms per milliliter (ng/mL)
    number analyzed (Participants) | 8 | 3 | 11
    (all) | 311.6 (241.0) | 289.0 (109.7) | 305.5 (207.8)
N-terminal propeptide of BNP (NT-proBNP) [Mean (Standard Deviation); unit: Nanograms per liter (ng/L)] — Biomarkers were determined in plasma/serum by a central laboratory using validated assays platforms including appropriate quality controls. Population: Participants in full analysis set (FAS) with evaluable data for this evaluation
  Nanograms per liter (ng/L)
    number analyzed (Participants) | 9 | 7 | 16
    (all) | 11972.4 (20747.7) | 2927.4 (3742.5) | 8015.3 (16020.7)
High sensitive Troponin T [Mean (Standard Deviation); unit: Picograms per millilitre (pg/mL)] — Biomarkers were determined in plasma/serum by a central laboratory using validated assays platforms including appropriate quality controls. Values below lower limit of quantification (LLOQ) were substituted by 1/2 LLOQ for the calculation of statistics (LLOQ = 13.0) Population: Participants in full analysis set (FAS) with evaluable data for this evaluation
  Picograms per millilitre (pg/mL)
    number analyzed (Participants) | 9 | 7 | 16
    (all) | 58.58 (46.30) | 22.73 (6.99) | 42.89 (38.74)
Blood pressure [Mean (Standard Deviation); unit: millimetre of mercury (mmHg)] — Systolic blood pressure (SBP) and diastolic blood pressure (DBP) were collected. Population: Participants in full analysis set (FAS) with evaluable data for this evaluation
  millimetre of mercury (mmHg)
    SBP: number analyzed (Participants) | 11 | 12 | 23
    SBP | 114.0 (17.6) | 124.0 (15.5) | 119.2 (16.9)
    DBP: number analyzed (Participants) | 11 | 12 | 23
    DBP | 69.3 (11.9) | 66.3 (12.0) | 67.7 (11.7)
Heart rate [Mean (Standard Deviation); unit: Beats per minute] — Population: Participants in full analysis set (FAS) with evaluable data for this evaluation
  Beats per minute
    number analyzed (Participants) | 11 | 12 | 23
    (all) | 69.5 (12.8) | 78.7 (17.0) | 74.3 (15.5)
Interventricular septal wall thickness [Mean (Standard Deviation); unit: Millimeters (mm)] — Interventricular septal wall thickness was measured by echocardiography. Population: Participants in full analysis set (FAS) with evaluable data for this evaluation
  Millimeters (mm)
    number analyzed (Participants) | 11 | 10 | 21
    (all) | 10.377 (3.178) | 11.974 (1.478) | 11.138 (2.589)
Diameter of the left ventricle in diastole [Mean (Standard Deviation); unit: Millimeters (mm)] — Diameter of the left ventricle in diastole was measured by echocardiography. Population: Participants in full analysis set (FAS) with evaluable data for this evaluation
  Millimeters (mm)
    number analyzed (Participants) | 13 | 10 | 23
    (all) | 64.085 (7.074) | 48.369 (6.001) | 57.252 (10.271)
Diameter of the left ventricle in systole [Mean (Standard Deviation); unit: Millimeters (mm)] — Diameter of the left ventricle in systole was measured by echocardiography. Population: Participants in full analysis set (FAS) with evaluable data for this evaluation
  Millimeters (mm)
    number analyzed (Participants) | 9 | 9 | 18
    (all) | 55.278 (7.119) | 32.778 (4.302) | 44.028 (12.906)
Left ventricular end-diastolic volume [Mean (Standard Deviation); unit: Milliliter (mL)] — Left ventricular end-diastolic volume was measured by echocardiography. Population: Participants in full analysis set (FAS) with evaluable data for this evaluation
  Milliliter (mL)
    number analyzed (Participants) | 10 | 7 | 17
    (all) | 224.480 (42.473) | 89.846 (27.972) | 169.042 (77.285)
Left ventricular end-systolic volume [Mean (Standard Deviation); unit: Milliliter (mL)] — Left ventricular end-systolic volume was measured by echocardiography. Population: Participants in full analysis set (FAS) with evaluable data for this evaluation
  Milliliter (mL)
    number analyzed (Participants) | 11 | 7 | 18
    (all) | 151.61 (32.46) | 41.49 (16.37) | 108.78 (61.37)
Left ventricular ejection fraction [Mean (Standard Deviation); unit: Percentage of the volumn of blood] — Left ventricular ejection fraction was measured by echocardiography. Population: Participants in full analysis set (FAS) with evaluable data for this evaluation
  Percentage of the volumn of blood
    number analyzed (Participants) | 13 | 10 | 23
    (all) | 28.54 (6.83) | 53.56 (5.58) | 39.42 (14.11)
Left atrial end-systolic volume [Mean (Standard Deviation); unit: Milliliter (mL)] — Left atrial end-systolic volume was measured by echocardiography. Population: Participants in full analysis set (FAS) with evaluable data for this evaluation
  Milliliter (mL)
    number analyzed (Participants) | 12 | 7 | 19
    (all) | 115.708 (56.175) | 86.517 (22.065) | 104.954 (47.959)
Left atrial end systolic volume index [Mean (Standard Deviation); unit: Milliliter per square meter (mL/m^2)] — Left atrial end systolic volume index was measured by echocardiography. Population: Participants in full analysis set (FAS) with evaluable data for this evaluation
  Milliliter per square meter (mL/m^2)
    number analyzed (Participants) | 12 | 7 | 19
    (all) | 60.4508 (33.8365) | 44.5747 (14.0789) | 54.6017 (28.7688)
Mitral peak velocity of late filling (A) [Mean (Standard Deviation); unit: Centimeter per second (cm/sec)] — Mitral peak velocity of late filling (A) was measured by echocardiography. Population: Participants in full analysis set (FAS) with evaluable data for this evaluation
  Centimeter per second (cm/sec)
    number analyzed (Participants) | 7 | 8 | 15
    (all) | 54.89 (33.64) | 76.69 (37.44) | 66.51 (36.23)
Mitral peak velocity of early filling (E) [Mean (Standard Deviation); unit: Centimeter per second (cm/sec)] — Mitral peak velocity of early filling (E) was measured by echocardiography. Population: Participants in full analysis set (FAS) with evaluable data for this evaluation
  Centimeter per second (cm/sec)
    number analyzed (Participants) | 8 | 10 | 18
    (all) | 86.98 (40.43) | 65.56 (26.50) | 75.08 (34.13)
Mitral lateral annulus early diastolic peak velocity [Mean (Standard Deviation); unit: Centimeter per second (cm/sec)] — Mitral lateral annulus early diastolic peak velocity was measured by echocardiography. Population: Participants in full analysis set (FAS) with evaluable data for this evaluation
  Centimeter per second (cm/sec)
    number analyzed (Participants) | 8 | 8 | 16
    (all) | 8.899 (3.634) | 9.114 (2.991) | 9.006 (3.217)
Mitral septal annulus early diastolic peak velocity [Mean (Standard Deviation); unit: Centimeter per second (cm/sec)] — Mitral septal annulus early diastolic peak velocity was measured by echocardiography. Population: Participants in full analysis set (FAS) with evaluable data for this evaluation
  Centimeter per second (cm/sec)
    number analyzed (Participants) | 8 | 8 | 16
    (all) | 4.949 (2.229) | 12.139 (15.744) | 8.544 (11.479)
Tricuspid annular plane systolic excursion [Mean (Standard Deviation); unit: Millimeters (mm)] — Tricuspid annular plane systolic excursion was measured by echocardiography. Population: Participants in full analysis set (FAS) with evaluable data for this evaluation
  Millimeters (mm)
    number analyzed (Participants) | 13 | 11 | 24
    (all) | 16.612 (3.734) | 18.295 (6.178) | 17.383 (4.960)
Pressure gradient of tricuspid valve [Mean (Standard Deviation); unit: Millimetre of mercury (mmHg)] — Pressure gradient of tricuspid valve was measured by echocardiography. Population: Participants in full analysis set (FAS) with evaluable data for this evaluation
  Millimetre of mercury (mmHg)
    number analyzed (Participants) | 12 | 9 | 21
    (all) | 40.937 (19.458) | 53.038 (32.335) | 46.123 (25.771)
Right atrial mean pressure [Mean (Standard Deviation); unit: Millimetre of mercury (mmHg)] — Right atrial mean pressure was measured by echocardiography. Population: Participants in full analysis set (FAS) with evaluable data for this evaluation
  Millimetre of mercury (mmHg)
    number analyzed (Participants) | 10 | 9 | 19
    (all) | 8.8 (5.7) | 5.4 (4.2) | 7.2 (5.2)
Number of participants per NYHA classification [Count of Participants; unit: Participants] — New York Heart Association (NYHA) Classification: Class I = No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc. Class II = Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity. Class III = Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m). Comfortable only at rest. Class IV = Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients. Population: Participants in full analysis set (FAS) with evaluable data for this evaluation
  Participants
    number analyzed (Participants) | 13 | 12 | 25
    NYHA Class II | 6 | 2 | 8
    NYHA Class III | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: Daily Steps Count
Description: Daily steps count was measured with DynaPort Move Monitor device and evaluated to reflect the amount of daily physical activity.
Time Frame: At Day 9 and Day 77
Population: Device set (DES): All participants with DynaPort parameters for least one wearing period
Measure: Mean (Standard Deviation); unit: Steps
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 7 | 8
Steps
  Day 9: number analyzed (Participants) | 7 | 6
  Day 9 | 5052 (3090) | 3509 (1871)
  Day 77: number analyzed (Participants) | 4 | 8
  Day 77 | 6627 (3851) | 2524 (1606)

2. Primary Outcome: Daily Physical Activity Level
Description: Movement intensity of an activity, which was the average body acceleration (g) during this activity, was measured with DynaPort Move Monitor device and evaluated as daily physical activity level (PAL). Higher values indicate higher physical activity level and intensity.
Time Frame: At Day 9 and Day 77
Population: Device set (DES): All participants with DynaPort parameters for least one wearing period
Measure: Mean (Standard Deviation); unit: Meter*second^-2 (m*s^-2)
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 7 | 8
Meter*second^-2 (m*s^-2)
  Day 9: number analyzed (Participants) | 7 | 6
  Day 9 | 1.612 (0.135) | 1.606 (0.138)
  Day 77: number analyzed (Participants) | 4 | 8
  Day 77 | 1.678 (0.153) | 1.586 (0.144)

3. Primary Outcome: Total Daily Energy Expenditure
Description: Total daily energy expenditure was measured with DynaPort Move Monitor device and evaluated to reflect the amount of daily physical activity.
Time Frame: At Day 9 and Day 77
Population: Device set (DES): All participants with DynaPort parameters for least one wearing period
Measure: Mean (Standard Deviation); unit: Kilocalorie (kcal)
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 7 | 8
Kilocalorie (kcal)
  Day 9: number analyzed (Participants) | 7 | 6
  Day 9 | 2445 (378) | 2380 (557)
  Day 77: number analyzed (Participants) | 4 | 8
  Day 77 | 2374 (322) | 2329 (494)

4. Primary Outcome: Duration of Daily Physical Activity
Description: Duration of daily physical activity was measured with DynaPort Move Monitor device.
Time Frame: At Day 9 and Day 77
Population: Device set (DES): All participants with DynaPort parameters for least one wearing period
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 7 | 8
Hours
  Active Time - Day 9: number analyzed (Participants) | 7 | 6
  Active Time - Day 9 | 4.157 (1.631) | 3.843 (1.886)
  Active Time - Day 77: number analyzed (Participants) | 4 | 8
  Active Time - Day 77 | 5.043 (1.578) | 3.861 (2.796)

5. Primary Outcome: Time Duration Per Activity Status
Description: Time duration per activity status was measured with DynaPort Move Monitor device and evaluated to reflect the intensity of daily physical activity. Physical Activity intensities use absolute aerobic intensity in terms of Metabolic Equivalent of Task (MET), which is a physiological concept expressing the energy cost of a physical activity as a multiple of Basal Metabolic Rate (BMR). By convention, 1 MET is considered as the resting metabolic rate obtained during quiet sitting. According to the American College of Sports Medicine (ACSM) thresholds for adults: Light-intensity activities are defined as 1.1 MET to 2.9 METs; Moderate-intensity activities are defined as 3.0 to 5.9 METs; Vigorous-intensity activities are defined as 6.0 METs or more.
Time Frame: At Day 9 and Day 77
Population: Device set (DES): All participants with DynaPort parameters for least one wearing period
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 7 | 8
Hours
  Time in Sedentary State - Day 9: number analyzed (Participants) | 7 | 6
  Time in Sedentary State - Day 9 | 20.957 (1.180) | 21.196 (1.346)
  Time in Sedentary State - Day 77: number analyzed (Participants) | 4 | 8
  Time in Sedentary State - Day 77 | 20.415 (1.457) | 21.203 (1.402)
  Time in Light Activity State - Day 9: number analyzed (Participants) | 7 | 6
  Time in Light Activity State - Day 9 | 1.156 (0.632) | 1.275 (0.779)
  Time in Light Activity State - Day 77: number analyzed (Participants) | 4 | 8
  Time in Light Activity State - Day 77 | 1.586 (0.723) | 1.415 (1.043)
  Time in Moderate Activity State - Day 9: number analyzed (Participants) | 7 | 6
  Time in Moderate Activity State - Day 9 | 1.365 (0.515) | 1.194 (0.459)
  Time in Moderate Activity State - Day 77: number analyzed (Participants) | 4 | 8
  Time in Moderate Activity State - Day 77 | 1.471 (0.397) | 0.995 (0.500)
  Time in Vigorous Activity State - Day 9: number analyzed (Participants) | 7 | 6
  Time in Vigorous Activity State - Day 9 | 0.181 (0.355) | 0.033 (0.036)
  Time in Vigorous Activity State - Day 77: number analyzed (Participants) | 4 | 8
  Time in Vigorous Activity State - Day 77 | 0.357 (0.562) | 0.019 (0.022)

6. Secondary Outcome: 6-minute Walking Distance (6MWD)
Description: 6-minute walking distance (6MWD) is a exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. An increase in the distance walked indicates improvement in basic mobility.
Time Frame: At Day 84
Population: Participants in full analysis set (FAS, all participants that were enrolled into the study and that wore at least one device) with evaluable data for this assessment
Measure: Mean (Full Range); unit: Meters
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 9 | 10
Meters | 456 [251 to 828] | 261 [92 to 414]

7. Secondary Outcome: Sleep Movements
Description: Sleep movements was measured with DynaPort Move Monitor device.
Time Frame: Up to Day 84
Population: No participant in device set (DES) with evaluable data for this evaluation
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Sleep Patterns
Description: Sleep patterns was measured with DynaPort Move Monitor device.
Time Frame: Up to Day 84
Population: No participant in device set (DES) with evaluable data for this evaluation
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Sit-to-stand Behaviour
Description: Sit-to-stand behaviour was measured with DynaPort Move Monitor device.
Time Frame: Up to Day 84
Population: No participant in device set (DES) with evaluable data for this evaluation
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Quality of Life as Measured With the Kansas City Cardiomyopathy Questionnaire Score
Description: The Kansas City Cardiomyopathy Questionnaire (KCCQ) is the leading health-related quality-of-life measure for patients with heart failure (HF). It is a 23-item questionnaire that independently measures the impact of patients' HF, or its treatment, on 7 distinct domains: symptom frequency, symptom burden, physical limitation, quality of life, social limitations, self-efficacy and symptoms stability. Physical Limitation ranges 0-100. Total Symptom Score (range 0-100) combines the Symptom Frequency and the Symptom Burden scores; Clinical Summary Score (range 0-100) combines the Total Symptom and Physical Limitation scores to replicate the NYHA classification; Overall Summary Score (range 0-100) includes the Total Symptom, Physical Limitation, Social Limitations, and Quality of Life scores. Higher scores indicate more favorable states.
Time Frame: At Day 9 and Day 84
Population: Participants in full analysis set (FAS, all participants that were enrolled into the study and that wore at least one device) with evaluable data on each evaluation day for this assessment
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 12 | 12
Scores on a scale
  Total Symptom Score - Day 9: number analyzed (Participants) | 7 | 6
  Total Symptom Score - Day 9 | 75.0 [48 to 100] | 48.5 [0 to 71]
  Total Symptom Score - Day 84: number analyzed (Participants) | 5 | 6
  Total Symptom Score - Day 84 | 75.0 [55 to 100] | 39.5 [2 to 65]
  Clinical Summary Score - Day 9: number analyzed (Participants) | 7 | 6
  Clinical Summary Score - Day 9 | 69.0 [45 to 100] | 40.0 [3 to 56]
  Clinical Summary Score - Day 84: number analyzed (Participants) | 5 | 6
  Clinical Summary Score - Day 84 | 67.0 [52 to 100] | 36.0 [9 to 48]
  Overall Summary Score - Day 9: number analyzed (Participants) | 7 | 6
  Overall Summary Score - Day 9 | 57.0 [38 to 92] | 39.5 [2 to 70]
  Overall Summary Score - Day 84: number analyzed (Participants) | 5 | 6
  Overall Summary Score - Day 84 | 62.0 [42 to 100] | 36.5 [6 to 51]
  Physical Limitation Score - Day 9: number analyzed (Participants) | 6 | 6
  Physical Limitation Score - Day 9 | 71.0 [42 to 79] | 34.0 [6 to 46]
  Physical Limitation Score - Day 84: number analyzed (Participants) | 4 | 6
  Physical Limitation Score - Day 84 | 73.0 [29 to 100] | 28.0 [13 to 38]

11. Secondary Outcome: Quality of Life as Measured With the PRO - Activity Scores
Description: REALIsM-HF exploratory daily questionnaire was developed to include patient-reported outcome (PRO) items that can be administered as a daily diary in the study. Overall activity score ranges from 0 to 240 and general physical activity score ranges from 0 to 4. Higher scores indicate more favorable states.
Time Frame: At Day 9 and Day 77
Population: as for outcome 10
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 11 | 10
Scores on a scale
  Overall Activity Score - Day 9: number analyzed (Participants) | 7 | 6
  Overall Activity Score - Day 9 | 75.909 [49.89 to 198.08] | 107.708 [70.00 to 145.17]
  Overall Activity Score - Day 77: number analyzed (Participants) | 4 | 4
  Overall Activity Score - Day 77 | 108.486 [27.73 to 224.00] | 106.700 [86.75 to 121.93]
  General Physical Activity Score - Day 9: number analyzed (Participants) | 7 | 6
  General Physical Activity Score - Day 9 | 1.70000 [0.8889 to 2.3333] | 1.66667 [0.7500 to 2.7778]
  General Physical Activity Score - Day 77: number analyzed (Participants) | 4 | 4
  General Physical Activity Score - Day 77 | 1.48413 [0.3636 to 2.5556] | 1.53333 [1.2500 to 1.70000]

12. Secondary Outcome: Quality of Life as Measured With the PRO - Change in Activities and Symptoms
Description: REALIsM-HF exploratory daily questionnaire was developed to include patient-reported outcome (PRO) items that can be administered as a daily diary in the study. Answers to question "How have your physical activities changed since you were discharged from the hospital": 1= Very much more physically active; 2= Much more physically active; 3= A little more physically active; 4= No change in physical activities; 5= A little less physically active; 6= Much less physically active; 7= Very much less physically active. Answers to questions "How has your feeling of tiredness changed since you were discharged from the hospital", "How has your shortness of breath changed since you were discharged from the hospital" and "How has your swelling in your legs, ankles, or feet changed since you were discharged from the hospital": 1= Very much improved; 2= Much improved; 3= Minimally improved; 4= No change; 5= Minimally worse; 6= Much worse; 7= Very much worse.
Time Frame: At Day 9 and Day 77
Population: as for outcome 10
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 11 | 10
Scores on a scale
  How Have Your Physical Activities Changed Since Discharged from Hospital - Day 9: number analyzed (Participants) | 7 | 6
  How Have Your Physical Activities Changed Since Discharged from Hospital - Day 9 | 2.0 [2 to 6] | 4.0 [3 to 7]
  How Have Your Physical Activities Changed Since Discharged from Hospital - Day 77: number analyzed (Participants) | 5 | 6
  How Have Your Physical Activities Changed Since Discharged from Hospital - Day 77 | 3.0 [2 to 6] | 4.5 [3 to 7]
  How Has Your Feeling of Tiredness Changed Since Discharged from Hospital - Day 9: number analyzed (Participants) | 7 | 6
  How Has Your Feeling of Tiredness Changed Since Discharged from Hospital - Day 9 | 2.0 [2 to 4] | 4.5 [3 to 7]
  How Has Your Feeling of Tiredness Changed Since Discharged from Hospital - Day 77: number analyzed (Participants) | 5 | 6
  How Has Your Feeling of Tiredness Changed Since Discharged from Hospital - Day 77 | 2.0 [2 to 4] | 4.0 [2 to 6]
  How Has Your Shortness of Breath Changed Since Discharged from Hospital - Day 9: number analyzed (Participants) | 7 | 6
  How Has Your Shortness of Breath Changed Since Discharged from Hospital - Day 9 | 2.0 [1 to 6] | 4.0 [3 to 6]
  How Has Your Shortness of Breath Changed Since Discharged from Hospital - Day 77: number analyzed (Participants) | 5 | 6
  How Has Your Shortness of Breath Changed Since Discharged from Hospital - Day 77 | 2.0 [2 to 6] | 4.5 [3 to 7]
  How Has Your Swelling in Your Legs, Ankles, or Feet Changed Since Discharged from Hospital - Day 9: number analyzed (Participants) | 7 | 6
  How Has Your Swelling in Your Legs, Ankles, or Feet Changed Since Discharged from Hospital - Day 9 | 4.0 [1 to 4] | 3.5 [2 to 7]
  How Has Your Swelling in Your Legs, Ankles, or Feet Changed Since Discharged from Hospital - Day 77: number analyzed (Participants) | 5 | 6
  How Has Your Swelling in Your Legs, Ankles, or Feet Changed Since Discharged from Hospital - Day 77 | 2.0 [2 to 4] | 4.0 [3 to 6]

13. Secondary Outcome: Copeptin
Description: Blood sample for biomarkers including Copeptin were collected from participants in order to validate such biomarkers for clinical use in the context of heart failure. Biomarkers concentration was determined in plasma/serum by a central laboratory using validated assays platforms including appropriate quality controls.
Time Frame: At Day 9 and Day 84
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Picomoles per litre (pmol/L)
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 14 | 13
Picomoles per litre (pmol/L)
  Day 9: number analyzed (Participants) | 8 | 7
  Day 9 | 41.553 (36.802) | 29.457 (25.633)
  Day 84: number analyzed (Participants) | 9 | 11
  Day 84 | 31.743 (19.022) | 34.221 (23.304)

14. Secondary Outcome: Galectin-3
Description: Blood sample for biomarkers including Galectin-3 were collected from participants in order to validate such biomarkers for clinical use in the context of heart failure. Biomarkers concentration was determined in plasma/serum by a central laboratory using validated assays platforms including appropriate quality controls.
Time Frame: At Day 9 and Day 84
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 14 | 13
Nanograms per milliliter (ng/mL)
  Day 9: number analyzed (Participants) | 8 | 7
  Day 9 | 16.736 (10.883) | 14.461 (6.036)
  Day 84: number analyzed (Participants) | 9 | 11
  Day 84 | 12.637 (8.082) | 17.947 (14.908)

15. Secondary Outcome: Growth Differentiation Factor 15 (GDF 15)
Description: Blood sample for biomarkers including GDF 15 were collected from participants in order to validate such biomarkers for clinical use in the context of heart failure. Biomarkers concentration was determined in plasma/serum by a central laboratory using validated assays platforms including appropriate quality controls.
Time Frame: At Day 9 and Day 84
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Picograms per millilitre (pg/mL)
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 14 | 13
Picograms per millilitre (pg/mL)
  Day 9: number analyzed (Participants) | 8 | 7
  Day 9 | 5297.4 (6452.6) | 1987.7 (913.7)
  Day 84: number analyzed (Participants) | 9 | 11
  Day 84 | 2796.8 (1942.1) | 2333.3 (1497.8)

16. Secondary Outcome: Human Interleukin-1 Receptor 4 / ST2 (sST2)
Description: Blood sample for biomarkers including sST2 were collected from participants in order to validate such biomarkers for clinical use in the context of heart failure. Biomarkers concentration was determined in plasma/serum by a central laboratory using validated assays platforms including appropriate quality controls. Values above upper limit of quantification (ULOQ) were substituted by ULOQ for the calculation of statistics (ULOQ = 80.0)
Time Frame: At Day 9 and Day 84
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Picograms per litre (pg/L)
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 14 | 13
Picograms per litre (pg/L)
  Day 9: number analyzed (Participants) | 8 | 7
  Day 9 | 34.88 (13.63) | 23.27 (8.45)
  Day 84: number analyzed (Participants) | 9 | 11
  Day 84 | 26.13 (21.51) | 24.35 (9.98)

17. Secondary Outcome: Human Insulin-like Growth Factor Binding (IGFBP7)
Description: Blood sample for biomarkers including IGFBP7 were collected from participants in order to validate such biomarkers for clinical use in the context of heart failure. Biomarkers concentration was determined in plasma/serum by a central laboratory using validated assays platforms including appropriate quality controls.
Time Frame: At Day 9 and Day 84
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 13 | 10
Nanograms per milliliter (ng/mL)
  Day 9: number analyzed (Participants) | 8 | 6
  Day 9 | 293.9 (156.4) | 256.5 (112.8)
  Day 84: number analyzed (Participants) | 5 | 4
  Day 84 | 228.8 (49.5) | 242.5 (98.8)

18. Secondary Outcome: N-terminal Propeptide of BNP (NT-proBNP)
Description: Blood sample for biomarkers including NT-proBNP were collected from participants in order to validate such biomarkers for clinical use in the context of heart failure. Biomarkers concentration was determined in plasma/serum by a central laboratory using validated assays platforms including appropriate quality controls.
Time Frame: At Day 9 and Day 84
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Nanograms per liter (ng/L)
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 14 | 13
Nanograms per liter (ng/L)
  Day 9: number analyzed (Participants) | 8 | 7
  Day 9 | 10985.4 (22390.8) | 2051.7 (2434.9)
  Day 84: number analyzed (Participants) | 9 | 9
  Day 84 | 3660.0 (3463.7) | 2746.6 (3395.6)

19. Secondary Outcome: High Sensitive Troponin T (hsTRT)
Description: Blood sample for biomarkers including hsTRT were collected from participants in order to validate such biomarkers for clinical use in the context of heart failure. Biomarkers concentration was determined in plasma/serum by a central laboratory using validated assays platforms including appropriate quality controls. Values below lower limit of quantification (LLOQ) were substituted by 1/2 LLOQ for the calculation of statistics (LLOQ = 13.0)
Time Frame: At Day 9 and Day 84
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Picograms per millilitre (pg/mL)
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 14 | 13
Picograms per millilitre (pg/mL)
  Day 9: number analyzed (Participants) | 8 | 7
  Day 9 | 46.56 (35.00) | 24.70 (5.98)
  Day 84: number analyzed (Participants) | 9 | 10
  Day 84 | 33.82 (25.85) | 27.00 (8.40)

20. Secondary Outcome: Blood Pressure
Description: Systolic blood pressure (SBP) and diastolic blood pressure (DBP) were collected.
Time Frame: At Day 9, Day 77 and Day 84
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: millimetre of mercury (mmHg)
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 14 | 13
millimetre of mercury (mmHg)
  SBP - Day 9: number analyzed (Participants) | 11 | 13
  SBP - Day 9 | 108.1 (14.6) | 128.8 (18.6)
  SBP - Day 77: number analyzed (Participants) | 8 | 11
  SBP - Day 77 | 114.1 (27.7) | 126.6 (14.5)
  SBP - Day 84: number analyzed (Participants) | 9 | 11
  SBP - Day 84 | 117.6 (15.2) | 124.5 (12.5)
  DBP - Day 9: number analyzed (Participants) | 11 | 13
  DBP - Day 9 | 66.3 (10.7) | 72.7 (14.6)
  DBP - Day 77: number analyzed (Participants) | 8 | 11
  DBP - Day 77 | 63.9 (14.6) | 64.5 (12.8)
  DBP - Day 84: number analyzed (Participants) | 9 | 11
  DBP - Day 84 | 70.0 (12.2) | 65.1 (13.0)

21. Secondary Outcome: Heart Rate
Description: Heart rate data were collected by electrocardiogram (ECG).
Time Frame: At Day 9, Day 77 and Day 84
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 14 | 13
Beats per minute
  Day 9: number analyzed (Participants) | 11 | 13
  Day 9 | 68.0 (13.7) | 73.6 (18.0)
  Day 77: number analyzed (Participants) | 8 | 11
  Day 77 | 63.3 (15.2) | 70.3 (17.2)
  Day 84: number analyzed (Participants) | 9 | 11
  Day 84 | 68.0 (16.4) | 73.3 (20.2)

22. Secondary Outcome: Interventricular Septal Wall Thickness
Description: Interventricular septal wall thickness was measured by echocardiography.
Time Frame: At Day 84
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimeters (mm)
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 6 | 6
Millimeters (mm) | 13.317 (4.667) | 12.578 (0.899)

23. Secondary Outcome: Diameter of the Left Ventricle in Diastole
Description: Diameter of the left ventricle in diastole was measured by echocardiography.
Time Frame: At Day 84
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimeters (mm)
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 6 | 6
Millimeters (mm) | 64.465 (12.425) | 47.705 (4.003)

24. Secondary Outcome: Diameter of the Left Ventricle in Systole
Description: Diameter of the left ventricle in systole was measured by echocardiography.
Time Frame: At Day 84
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimeters (mm)
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 5 | 6
Millimeters (mm) | 53.318 (13.067) | 35.133 (5.369)

25. Secondary Outcome: Left Ventricular End-diastolic Volume
Description: Left ventricular end-diastolic volume was measured by echocardiography.
Time Frame: At Day 84
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Milliliter (mL)
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 6 | 5
Milliliter (mL) | 219.667 (83.868) | 97.000 (23.130)

26. Secondary Outcome: Left Ventricular End-systolic Volume
Description: Left ventricular end-systolic volume was measured by echocardiography.
Time Frame: At Day 84
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Milliliter (mL)
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 6 | 5
Milliliter (mL) | 154.83 (66.02) | 51.60 (29.10)

27. Secondary Outcome: Left Ventricular Ejection Fraction
Description: Left ventricular ejection fraction was measured by echocardiography.
Time Frame: At Day 84
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percentage of the volume of blood
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 6 | 5
Percentage of the volume of blood | 28.33 (10.97) | 48.80 (15.91)

28. Secondary Outcome: Left Atrial End-systolic Volume
Description: Left atrial end-systolic volume was measured by echocardiography.
Time Frame: At Day 84
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Milliliter (mL)
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 5 | 6
Milliliter (mL) | 109.200 (30.310) | 76.833 (27.549)

29. Secondary Outcome: Left Atrial End Systolic Volume Index
Description: Left atrial end systolic volume index was measured by echocardiography.
Time Frame: At Day 84
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Milliliter per square meter (mL/m^2)
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 5 | 6
Milliliter per square meter (mL/m^2) | 55.6008 (17.9289) | 38.9653 (18.0952)

30. Secondary Outcome: Mitral Peak Velocity of Early Filling (E)
Description: Mitral peak velocity of early filling (E) was measured by echocardiography.
Time Frame: At Day 84
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Centimeter per second (cm/sec)
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 4 | 6
Centimeter per second (cm/sec) | 81.28 (40.45) | 78.53 (29.66)

31. Secondary Outcome: Mitral Peak Velocity of Late Filling (A)
Description: Mitral peak velocity of late filling (A) was measured by echocardiography.
Time Frame: At Day 84
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Centimeter per second (cm/sec)
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 4 | 4
Centimeter per second (cm/sec) | 64.43 (23.98) | 67.23 (29.77)

32. Secondary Outcome: Mitral Lateral Annulus Early Diastolic Peak Velocity
Description: Mitral lateral annulus early diastolic peak velocity was measured by echocardiography.
Time Frame: At Day 84
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Centimeter per second (cm/sec)
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 4 | 6
Centimeter per second (cm/sec) | 8.625 (2.266) | 8.623 (2.781)

33. Secondary Outcome: Mitral Septal Annulus Early Diastolic Peak Velocity
Description: Mitral septal annulus early diastolic peak velocity was measured by echocardiography.
Time Frame: At Day 84
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Centimeter per second (cm/sec)
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 4 | 6
Centimeter per second (cm/sec) | 7.418 (3.296) | 6.267 (2.555)

34. Secondary Outcome: Tricuspid Annular Plane Systolic Excursion
Description: Tricuspid annular plane systolic excursion was measured by echocardiography.
Time Frame: At Day 84
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimeters (mm)
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 6 | 6
Millimeters (mm) | 17.833 (2.483) | 19.000 (2.898)

35. Secondary Outcome: Pressure Gradient of Tricuspid Valve
Description: Pressure gradient of tricuspid valve was measured by echocardiography.
Time Frame: At Day 84
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimetre of mercury (mmHg)
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 6 | 6
Millimetre of mercury (mmHg) | 35.793 (15.524) | 30.982 (10.333)

36. Secondary Outcome: Right Atrial Mean Pressure
Description: Right atrial mean pressure was measured by echocardiography.
Time Frame: At Day 84
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimetre of mercury (mmHg)
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 4 | 6
Millimetre of mercury (mmHg) | 9.0 (6.9) | 5.8 (4.9)

37. Secondary Outcome: Heart Rate Variability (HRV) Derived From ECG
Description: Heart rate variability (HRV) derived from ECG were measured with AVIVO MPM and VitalPatch biosensor
Time Frame: Up to Day 84
Population: Due to non-compatibility of systems, data could not be derived from the VitalPatch biosensor at the time of report preparation.
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 0 | 0

38. Secondary Outcome: Number of Participants Per NYHA Classification by Visit
Description: The New York Heart Association (NYHA) Classification provides a simple way of classifying the extent of heart failure. The Stages of Heart Failure: Class I = No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc. Class II = Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity. Class III = Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20 - 100 m). Comfortable only at rest. Class IV = Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
Time Frame: At Day 9 and Day 84
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 14 | 13
Participants
  Day 9: number analyzed (Participants) | 11 | 13
  Day 9: NYHA CLASS I | 0 | 1
  Day 9: NYHA CLASS II | 9 | 4
  Day 9: NYHA CLASS III | 2 | 8
  Day 84: number analyzed (Participants) | 10 | 11
  Day 84: NYHA CLASS I | 2 | 1
  Day 84: NYHA CLASS II | 5 | 4
  Day 84: NYHA CLASS III | 3 | 6

39. Other Pre Specified Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence in a participant after providing written informed consent for participation in the study. An AE may or may not be temporally or causally associated with the use of a medicinal product. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly and another medical important serious event as judged by the investigator.
Time Frame: From signing the ICF until follow-up visit (up to 7 months)
Population: Full analysis set (FAS): All participants that were enrolled into the study and that wore at least one device
Measure: Count of Participants; unit: Participants
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 14 | 13
Participants
  Any AE | 9 | 10
  Any SAE | 5 | 3

40. Primary Outcome: Amount of Daily Physical Activity Measured With VitalPatch Biosensor
Description: Amount of daily physical activity was collected and measured with VitalPatch biosensor.
Time Frame: Up to Day 84
Population: as for outcome 37
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 0 | 0

41. Primary Outcome: Duration of Daily Physical Activity Measured With VitalPatch Biosensor
Description: Duration of daily physical activity was collected and measured with VitalPatch biosensor.
Time Frame: Up to Day 84
Population: as for outcome 37
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 0 | 0

42. Primary Outcome: Intensity of Daily Physical Activity Measured With VitalPatch Biosensor
Description: Intensity of daily physical activity was collected and measured with VitalPatch biosensor.
Time Frame: Up to Day 84
Population: as for outcome 37
Arm/Group | HFrEF | HFpEF
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From signing the informed consent form (ICF) until follow-up visit (up to 7 months)
Arm/Group | HFrEF | HFpEF
All-Cause Mortality (participants affected / at risk) | 1/14 | 1/13
Serious Adverse Events (participants affected / at risk) | 5/14 | 3/13
Other Adverse Events (participants affected / at risk) | 8/14 | 9/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HFrEF (N=14) | HFpEF (N=13)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia legionella (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Mitral valve repair (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HFrEF (N=14) | HFpEF (N=13)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0)
Tongue disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 3 (4)
Pain (General disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Catheterisation cardiac (Investigations) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Implantable defibrillator insertion (Surgical and medical procedures) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to non-compatibility of systems, data could not be derived from the VitalPatch biosensor at the time of report preparation. No evaluation was possible within this report. Further, activity data of the previous AVIVO patch as well as of the VitalPatch biosensor were not found to be scientifically evaluable. Activity data therefore were decided to be evaluated based on the DynaPort output only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-02-21): https://cdn.clinicaltrials.gov/large-docs/39/NCT03507439/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/39/NCT03507439/SAP_001.pdf